CLINICAL TRIAL: NCT03677427
Title: Randomized Trial Comparing 5 and 15 Fractions for Whole Breast Irradiation After Breast Conserving Surgery
Brief Title: Comparing 5 and 15 Fractions for Whole Breast Irradiation After Breast Conserving Surgery
Acronym: YO-HAI5
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Ghent (Other)
Collaborators: Kom Op Tegen Kanker (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EC/2017/0974 (BC-01085)
Record Dates: First submitted 2017-12-22; First posted 2018-09-19 (Actual); Last update posted 2024-03-05 (Actual); Status verified 2024-03

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Radiation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 5 fractions (Experimental)
  Interventions: Radiation: Radiation
- 15 fractions (Experimental)
  Interventions: Radiation: Radiation

INTERVENTIONS:
Radiation: Radiation — Radiation in breast cancer

SUMMARY:
Adjuvant radiotherapy after breast-conserving surgery for breast cancer reduces the risk of locoregional relapse and ensures better overall survival. In recent years it has been found that hypofractionation in which the number of radiation sessions is reduced with a higher dose per session offers advantages for breast irradiation. Randomized studies showed that moderate hypofraction regimens in 15 or 16 fractions have the same effect in tumor control and toxicity, although the total dose is lower than the traditional 50 Gy in 25 fractions. In a randomized study from the United Kingdom (START-B trial) even a better disease-free survival was seen with 15 sessions than with 25 sessions and the long-term side effects were also less with the short schedule.

This project proposes a clinical trial with an accelerated radiotherapy schedule in 5 sessions. It is expected that the accelerated schedule of 5 sessions over 12 days will have a number of radiobiological benefits: since a higher dose per session is given over a shorter period of time, it is expected that tumor control and survival will be higher. By reducing the total treatment time, the total dose is reduced, which may result in fewer radiation-related side effects and thus improve the quality of life. Apart from these radiobiological benefits, the shorter radiotherapy program reduces the number of treatment days from 15 to 5. This is not only more comfortable for the patients, but also increases the treatment capacity of the radiotherapy department. This opens up a possibility for the use of more complex techniques with fewer side effects such as radiation in the prone position.

This project includes a randomized study comparing the accelerated schedule in 5 sessions with a hypofraction schedule of 15 sessions in patients who are irradiated on the entire breast after breast-saving surgery. The primary endpoint is chest retraction (loss of volume) 2 years after radiotherapy.

DETAILED DESCRIPTION:
Adjuvant radiotherapy after breast conserving surgery for breast cancer reduces the locoregional recurrence rate and improves overall survival. In recent years, it has become clear that breast cancer cells are more sensitive to fraction dose than originally presumed. Large randomized trials confirm this hypothesis: moderate hypofractionation schemes in 15 or 16 fractions are at least equivalent in tumor control and toxicity although the total dose is lower than the traditional 50 Gy in 25 fractions. Further acceleration to 5 fractions is expected to have an even larger radiobiological advantage regarding tumor control. Additional advantages are patient comfort and a better use of radiotherapy resources. Due to capacity problems some radiotherapy departments are faced with waiting lists which not only delay the time between surgery and radiotherapy, but also interfere with the introduction of more sophisticated treatment techniques like prone whole-breast irradiation (WBI). Prone WBI has several advantages over supine WBI: less acute skin toxicity and improved breast cosmesis and reduced doses to heart and lung leading to less radiation-induced heart diseases and secondary lung cancer induction.

Hypofractionation and acceleration (shorter radiotherapy schemes with less fractions and a higher dose per fraction) are attractive both for the patient (less treatment sessions) and for the hospital (more treatment capacity and shorter waiting lists). Moderate hypofractionation in 15 or 16 fractions has been generally accepted as a valid alternative for the historical schedules of 25-30 fractions for whole-breast irradiation (WBI) after breast conserving surgery (BCS). With a median follow-up of 9.9 years, the UK START-B trial showed no significant difference in locoregional control between a hypofractionated schedule of 40.05 Gy in 15 fractions and a normofractionation scheme of 50 Gy in 25 fractions1. The Canadian schedule of 42.5 Gy in 16 fractions was also not inferior to the 50 Gy/25 fractions after 10 years of follow-up2. Aside from the obvious advantage of shortening the overall treatment time from 5 weeks to 3 weeks, both for the patient and the radiotherapy department, there might be some radiobiological advantages too. In the START-B trial, breast shrinkage, telangiectasia and breast oedema were significantly less frequent in the hypofractionation group. Better disease free survival and overall survival were also reported in the 15 fractions group, due to less distant relapses. The superiority of hypofractionation on survival and cosmesis was not observed in the Canadian trial.

While Belgium is a country with extensive health care facilities, some countries have a limited number of radiotherapy departments and patients have to travel a long distance for radiation. In those countries the pressure to evolve to even more retracted radiotherapy schemes is high. WBI in 5 fractions of 5.7 Gy over 5 weeks was tested in the FAST trial. A first analysis after 3 years demonstrated equivalence in toxicity and tumor control in comparison with the standard prescription of 25 x 2 Gy3. This accelerated schedule is in particular attractive for older patients since they often face logistic problems (frailty, impaired mobility, transportation difficulties). This sometimes leads to omission of radiotherapy leading to a reduced breast cancer specific survival4,5. For this reason, at UZ Gent a feasibility trial was started testing a highly accelerated schedule in 5 fractions over 12 days in patients of 65 years or older. The investigators used the FAST-scheme for WBI (5 x 5.7 Gy), but also included patients requiring a boost (5 x 6.5 Gy). With patient inclusion nearly finished, an interim analysis shows <10% grade 2-3 erythema, with only one case of moist desquamation, located at a skin fold6. In this study the investigators propose a multi-center randomized trial comparing our accelerated schedule in 5 fractions with a moderate hypofractionation scheme of 15 fractions in patients treated with WBI. The primary endpoint is breast retraction 2 years after radiotherapy.

ELIGIBILITY:
Inclusion Criteria:

* female patients with non-metastatic breast cancer,
* age ≥ 18 years,
* breast conserving surgery,
* multidisciplinary decision of adjuvant breast irradiation,
* informed consent obtained, signed and dated before specific protocol procedures

Exclusion Criteria:

* lymph node metastases,
* distant metastases,
* bilateral breast irradiation,
* history of previous radiation treatment to the same region
* life expectancy of less than 2 years,
* planned reconstructive surgery,
* conditions making toxicity evaluation difficult (e.g. skin disorders),
* inability to respect constraints on organs at risks
* patients unlikely to comply with the protocol

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — It's a study on breast cancer in female patients
Enrollment: 488 (Actual)
Dates: Start 2017-10-16 (Actual); Primary Completion 2023-06-23 (Actual); Study Completion 2023-06-23 (Actual)

PRIMARY OUTCOMES:
radiation-induced breast retraction | 4 years
  The primary endpoint of the randomized trial is radiation-induced breast retraction (volume loss) measured 2 years after radiotherapy.$

SECONDARY OUTCOMES:
Acute breast toxicity: dermatitis | 2 years
  Dermatitis, Common Terminology Criteria for Adverse Events v4.03
Acute breast toxicity: desquamation | 2 years
  Desquamation, Common Terminology Criteria for Adverse Events v4.03
Acute breast toxicity: breast oedema | 2 years
  Oedema, Common Terminology Criteria for Adverse Events v4.03
Acute breast toxicity: breast symptoms | 2 years
  pain, sense of heaviness, itching
Acute breast toxicity: dyspnoea | 2 years
  Dyspnoea, Common Terminology Criteria for Adverse Events v4.03
Acute breast toxicity: cough | 2 years
  Cough, Common Terminology Criteria for Adverse Events v4.03
Acute breast toxicity: pain | 2 years
  Pain, Common Terminology Criteria for Adverse Events v4.03
Late toxicity other than breast retraction: breast oedema | 5 years
  Breast oedema, Common Terminology Criteria for Adverse Events v4.03
Late toxicity other than breast retraction: telangiectasia | 5 years
  Telangiectasia, Late Effects Normal Tissue Task Force (LENT)-Subjective, Objective, Management, Analytic (SOMA) scales
Late toxicity other than breast retraction: colour changes | 5 years
  Colour changes, Common Terminology Criteria for Adverse Events v4.03
Late toxicity other than breast retraction: fibrosis | 5 years
  Fibrosis, Late Effects Normal Tissue Task Force (LENT)-Subjective, Objective, Management, Analytic (SOMA) scales
Late toxicity other than breast retraction: breast symptoms | 5 years
  Pain, sense of heaviness, itching
Late toxicity other than breast retraction: dyspnoe | 5 years
  Dyspnoe, Common Terminology Criteria for Adverse Events v4.03
Late toxicity other than breast retraction: pain | 5 years
  Pain, Common Terminology Criteria for Adverse Events v4.03

CONTACTS AND LOCATIONS:
Locations (1):
- Radiotherapie UZ Gent, Ghent, Oost-Vlaanderen, Belgium

IPD SHARING:
Plan to Share IPD: No